CLINICAL TRIAL: NCT01643291
Title: Ultrasound Imaging Facilitates Lumbar Punctures in Pediatric Oncology Patients With Difficult Surface Landmarks and/or a History of Difficult Lumbar Puncture
Brief Title: Ultrasound Use for Difficult Lumbar Punctures in Pediatric Oncology Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit subjects for this study.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tarun Bhalla, MD, Assistant Professor, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00335
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound (Experimental)
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound guidance for difficult lumbar punctures in the leukemic pediatric population.

SUMMARY:
Hematology-oncology patients may require frequent lumbar puncture for diagnosis, assessment and therapy. When LP is difficult, the patient may endure multiple attempts, prolonged anesthesia time, and with failure of LP may require fluoroscopy-guidance with associated radiation exposure. This investigation will evaluate lumbar punctures performed in the intraoperative setting by oncologists with ultrasound guidance performed by the anesthesiologist in the leukemic pediatric population. The investigators hypothesis is that anesthesiologist guided ultrasound assistance will decrease intraoperative time, number of attempts and need to have the procedure done with fluoroscopy minimizing radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing LP as per Heme-Onc clinic who have been deemed to be difficult LP placements.

Exclusion Criteria:

* Patients having concomitant procedures (bone marrow bx, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of punctures | 1 day
  Number of punctures required to obtain cerebral spinal fluid.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Ferre RM, Sweeney TW, Strout TD. Ultrasound identification of landmarks preceding lumbar puncture: a pilot study. Emerg Med J. 2009 Apr;26(4):276-7. doi: 10.1136/emj.2007.057455. PMID 19307389
- [Background] Abo A, Chen L, Johnston P, Santucci K. Positioning for lumbar puncture in children evaluated by bedside ultrasound. Pediatrics. 2010 May;125(5):e1149-53. doi: 10.1542/peds.2009-0646. Epub 2010 Apr 19. PMID 20403933
- [Background] Ayalin T, Lam SH. Ultrasound-assisted lumbar puncture in infants. Acad Emerg Med. 2011 Apr;18(4):e36. doi: 10.1111/j.1553-2712.2011.01044.x. No abstract available. PMID 21496132